CLINICAL TRIAL: NCT07245043
Title: The Effect of Sticker Intervention on Pain and Anxiety Experienced During IV Intervention
Brief Title: The Effect of Sticker Intervention on Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, HASRET YAĞMUR SEVİNÇ AKIN, Assistant Professor, Harran University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HRU/25.12.67
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: INTRAVENOUS CATHETER APPLICATION; Pain; Pain Management; Anxiety
Keywords: intravenous catheter application; children; pain management; anxiety
MeSH Terms: conditions — Pain; Agnosia; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Before implementing data collection tools, children and mothers will be informed, and data will be collected through face-to-face interviews using data collection forms after obtaining consent from those who agree to participate in the study. Children in the sticker group will be provided with stickers by the researcher during the application phase, which they can choose according to their own preferences.Children's anxiety and pain will be assessed based on both the researcher's and the child's reports before, during, and after the procedure, following consent from the mothers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sticker Group (Experimental): The researcher will provide stickers that children in the sticker group can choose according to their own preferences during the application phase.Children's anxiety and pain will be assessed based on both the researcher's and the child's reports before, during, and after the procedure, following consent from the mothers.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: control group — Children in the control group will not undergo any procedures other than routine hospital procedures. Children's anxiety and pain will be assessed based on both the researcher's and the child's reports before, during, and after the procedure, following consent from the mothers.

SUMMARY:
Peripheral venous catheterization, which involves the placement of an invasive device into the lumen of a peripheral vein, is a commonly used procedure in children receiving hospital treatment.IV insertion is a particularly painful and stressful experience for children. This is because children have more limited coping skills than adults. This study was designed as a randomized controlled trial to examine the effect of sticker intervention on pain and anxiety experienced during IV insertion.

DETAILED DESCRIPTION:
The study consists of an sticker group and a control group. Participants will be assigned to groups using stratified randomization. Anxiety levels in both groups will be assessed using the Children's Anxiety Scale-State (ÇAS-D), while pain levels will be evaluated by both the child and the researcher using a visual pain scale before, during, and after the procedure.For children in both groups, 10 minutes before the intravenous procedure, both the child and the researcher will rate the child's anxiety and pain using scales.During the IV procedure, the researcher will place the sticker chosen by the child on the IV insertion site. Meanwhile, the researcher will rate the child's anxiety and pain using scales. No sticker will be placed on the IV insertion site of the control group, and the child's anxiety and pain will be rated using scales.For both groups, 10 minutes after the intravenous procedure, both the child and the researcher will rate the child's anxiety and pain using scales.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-10 years,
* Children undergoing painful procedures
* Children undergoing IV procedures

Exclusion Criteria:

* Children who have undergone surgery,
* Children who have undergone procedures other than intravenous interventions,
* Children whose parents are not present,
* Children with any chronic illness or additional complaints that may trigger pain from the procedure,
* Children with mental retardation

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
1. Outcome Measures | For children in both groups: Ten minutes before the intravenous procedure, during the procedure, and ten minutes after the procedure, both the child and the researcher will rate the child's anxiety and pain using scales.
  The outcome measures for the sociodemographic data of the study will be collected using an "Information Form" containing questions about the child's age, gender, and descriptive characteristics such as whether they have previously had an intravenous catheter inserted.

OTHER OUTCOMES:
2. Outcome Measures | For children in both groups: Ten minutes before the intravenous procedure, during the procedure, and ten minutes after the procedure, both the child and the researcher will rate the child's pain using scales.
  Visual Pain Scale: The scale is a 10 cm line scaled from 1 to 10 to determine the severity of pain in children, with 10 representing maximum pain and 0 representing no pain. Patients are asked to mark a spot on the scale according to the pain they feel.
3. Outcome Measures | For children in both groups: Ten minutes before the intravenous procedure, during the procedure, and ten minutes after the procedure, both the child and the researcher will rate the child's anxiety using scales.
  Child Anxiety Scale-State (CAS-D): The scale is designed in the shape of a thermometer. Each horizontal line on the thermometer represents one point, and the light bulb at the bottom represents 0 points. As you move upward, the score increases, with a maximum of 10 points. A score of 0 on the scale indicates no anxiety, while a score of 10 indicates the highest level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: HASRET YAĞMUR SEVİNÇ AKIN, Assistant Professor, Study Director — Harran University; MAKSUDE YILDIRIM, Assistant Professor, Study Chair — Adiyaman University; BARIŞ AKIN, Specialist Nurse, Principal Investigator — MARDIN EDUCATION AND RESEARCH HOSPITAL
Locations (1):
- Mardin Education and Research Hospital, Mardin, Artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data from the study will be published as a scientific article.